CLINICAL TRIAL: NCT00338351
Title: To Assess Reactogenicity and Immunogenicity of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine, When Co-administered With GSK Biologicals' DTPa-HBV-IPV/Hib Vaccine (Infanrix™ Hexa) at 2, 4 and 6 Months of Age.
Brief Title: Safety and Immunogenicity Study of GlaxoSmithKline (GSK) Biologicals' 10-valent Pneumococcal Conjugate Vaccine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 106208
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: Pneumococcal (vaccine)

SUMMARY:
Three dose primary vaccination study of reactogenicity and immunogenicity in healthy infants between 6-12 weeks of age at the time of the first vaccination against Streptococcus pneumoniae.

DETAILED DESCRIPTION:
Test groups: 2 (120 subjects/group). 1 group receiving GSK Biologicals' 10-valent pneumococcal conjugate vaccine + DTPa combined vaccine; Control group receiving GSK Biologicals' Havrix + DTPa combined vaccine

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination, free of obvious health problems and with written informed consent obtained from the parent/guardian of the subject.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from one month before the first dose of vaccine(s) and during the entire study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240
Dates: Start 2006-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
After each dose: Grade 3 AEs

SECONDARY OUTCOMES:
After each dose: solicited/unsolicited AEs (4/31 days),SAEs (whole study); 1 month post 3: antibody concns to vaccine antigens

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lagos RE, Munoz AE, Levine MM, Lepetic A, Francois N, Yarzabal JP, Schuerman L. Safety and immunogenicity of the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Chilean children. Hum Vaccin. 2011 May;7(5):511-22. doi: 10.4161/hv.7.5.14634. Epub 2011 May 1. PMID 21441782
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 106208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106208 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register